CLINICAL TRIAL: NCT06376825
Title: The Efficacy and Acceptability of an Internet-Based Self-Help Program to Reduce Burnout Among Teachers: A Concurrent Multiple-Baseline Single-Case Experimental Study
Brief Title: The Efficacy and Acceptability of an Internet-Based Self-Help Program to Reduce Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Nalbant (Other)
Responsible Party: Sponsor-Investigator, Ahmet Nalbant, Psychiatrist, Researcher, CanSagligi Foundation
Organization: CanSagligi Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSV202401
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burnout, Professional
Keywords: Burnout; Acceptance and Commitment Therapy; İnternet-based psychotherapy; Single-case design
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The study will be a concurrent multiple-baseline single-case experimental study with participiants randomized to baseline durations.
Masking Description: In this study participants will be randomized to different baseline durations and randomization will be done by one of the investigators who are blind to participants assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MyLife Group (Experimental): In this concurrent multiple-baseline single-case experimental study, participants will have seven to fifteen days of baseline measurement with randomization.
  Interventions: Behavioral: MyLife: An internet-based self-help program to reduce burnout

INTERVENTIONS:
Behavioral: MyLife: An internet-based self-help program to reduce burnout — MyLife is a internet-based and Acceptance and Commitment Therapy oriented self-help program to reduce burnout. In this study a tailored to teachers version of the program will be used.

SUMMARY:
The goal of this clinical trial is to determine whether an internet-based self-help program reduces burnout in teachers. The study will also evaluate the program's acceptability which means assessing the extent to which users complete the program and find it useful. The main questions it aims to answer are:

* Does the program reduce the level of burnout in teachers?
* Does the program contribute to an increased sense of meaning for teachers?
* How much of the program do teachers finish?

DETAILED DESCRIPTION:
This concurrent multiple-baseline single-case experimental study aims to assess the efficacy and acceptability of an internet-based self-help program designed to mitigate burnout among teachers. The self-help program, named MyLife, adopts an Acceptance and Commitment Therapy framework and comprises eight modules. Preceding the commencement of the study, the program was tailored to address the specific needs of teachers through collaboration with people with lived experiences and the administration of nationwide surveys. Additionally, the daily questions utilized in this single-case study design were meticulously crafted for this study. In this study no guidance other than reminders will be offered.

Participants will be instructed to:

* Engage with program content, including audio and text components, every three days over a four-week period.
* Respond to daily questions once in day for eight weeks and both before and after the study, utilizing scales and questionnaires.

The research questions are as follows:

1. To what extent does the program alleviate burnout among teachers?
2. Does the program foster a heightened sense of meaning in teachers' professional lives?
3. What is the completion rate of the program among participating teachers?
4. Does the program effectively diminish experiential avoidance?

Hypotheses:

1. Teachers participating in the MyLife program will experience a significant decrease in burnout levels compared to baseline measures.
2. The MyLife program will lead to a significant increase in the perception of meaning in teachers' professional lives.
3. MyLife program will have a good acceptability.
4. Participation in the MyLife program will be associated with a significant reduction in experiential avoidance among teachers.

ELIGIBILITY:
Inclusion Criteria:

* Being a teacher in Türkiye
* Having burnout symptoms related to the workplace.
* Able to use e-mail, internet and mobile phone
* Able to read fluently in Turkish

Exclusion Criteria:

* Currently prescribed psychotropic medication or any change in psychotropic medication in last two months
* Currently undergoing psychotherapy.
* Having thoughts of suicide or self-mutilation.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Burnout Assessment Tool | At baseline and after 8 weeks
  Burnout Assessment Tool is a validated measure which evaluates to what extend people experience burnout in work place. The scale is a 5-point Likert type, meaning "1 = Never" to "5 = Always" (minimum:34 to maxiumum:150). Higher scores from the scale represent higher burnout. Turkish validity and reliability study was conducted and Cronbach's alpha value was stated as 0.95.
Valued Living Questionnaire | At baseline and after 8 weeks
  Valued Living Questionnaire is a validated measure and its aim is to evaluate valued living. The scale consists of 10 items with a 7-point Likert type as 0 = Not at all true and 6 = Completely true (minimum:0; maxiumum:60). The scale, for which Turkish validity and reliability studies have been conducted, has two sub-dimensions: "progress" and "blockage". While the progress subscale expresses that the person takes action in line with his values, the blockage dimension means that the person avoids certain experiences and moves away from a value-oriented life. The Cronbach's alpha value of the Turkish version of the scale was found to be 0.78; as for the progress sub-dimension was 0.77, and for the blockage dimension was 0.76.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire-2 | At baseline and after 8 weeks
  AAQ-2 is a measure aiming to evaluate experiential avoidance. The scale consists of 7-point Likert type (minimum:7 to maxiumum 49). Higher points indicate higher experiential avoidance.
System Usability Scale | After eight weeks
  System Usability Scale aims to measure evaluations of participants about an internet based program. It has 10 items which consists of 5-point Likert-type questions. Higher points indicate better usability of the system (Minimum:0 to maximum:100).
Attendance rate | After eight weeks.
  To evaluate acceptability, participants attendance rate to the program will be recorded.

OTHER OUTCOMES:
Daily measures | Daily questions will be asked during 8 weeks and data will be collected daily.
  Daily measures will include questions about burnout, valued living and experiential avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Nalbant, MD, Principal Investigator — CanSagligi Foundation Center for Contextual Behavioral Science
Locations (1):
- CanSagligi Foundation Center for Contextual Behavioral Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing would be available upon request